CLINICAL TRIAL: NCT00831272
Title: Pharmacogenetic Response to Naltrexone for Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Oslin (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, David Oslin, Sponsor-Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807991; 5R01AA017164-05 (NIH)
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): 50mg/day of naltrexone
  Interventions: Drug: naltrexone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: naltrexone — 50mg/day
  Other Names: ReVia
  Arms: Naltrexone
Drug: Placebo — Placebo
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The aims of the study are to test for treatment outcome differences in alcohol dependent subjects randomly assigned to 12 weeks of treatment with NTX (50mg/day) or placebo among those with one or two copies of the Asp40 allele of the mu-opioid receptor compared to those homozygous for the Asn40 allele. Thus, the design of the study is a 2X2 cell double-blind randomization to NTX or placebo stratified by genotype. To meet these aims, 150 alcohol dependent outpatients with one or two copies of the Asp40 variant of the mu-opioid receptor and 190 subjects homozygous for the Asn40 variant will be recruited across the four participating sites.

DETAILED DESCRIPTION:
Despite the well established efficacy of naltrexone, there are significant variations in individual responses to naltrexone. A critical question remains: under what circumstances and for which patients will naltrexone (NTX) be most beneficial? Recent work at our center provides evidence that the mu-opioid receptor (OPRM1) gene polymorphism A118G (Asn40Asp) imparts a significant change in treatment response. We have shown that patients with 1-2 copies of the Asp40 variant have significantly better treatment responses than patients with Asn40 variant (absence of heavy drinking -73.9% v/s 49% response). To further consolidate our knowledge, we wish to test the relationship between A118G polymorphism and the response to treatment with naltrexone. This work is focused on subjects of European or Asian descent as the A118G polymorphism occurs in less than 1% of those of African descent.

The study consists of 12 weeks of outpatient treatment with 50mg/day of naltrexone or placebo. Up to 340 subjects will be recruited across four sites. The inclusion criteria include adult males and females of European or Asian descent with DSM-IV diagnosis of alcohol dependence and heavy drinking per TLFB criteria. Patients with major psychiatric disorders or on psychotropic medications, other substance dependence problems (except nicotine), severe cognitive impairment, active suicidal/homicidal thoughts and serious medical conditions (including liver disorders) will be excluded.

The ultimate aim of this line of investigation is to further establish a genetic link between alcohol dependence and treatment by defining an endophenotype associated with treatment response.

Based upon these very promising findings, the aim of this study is to examine prospectively the interaction between a functional polymorphism of the mu-opioid receptor (A+118G (Asn40Asp)) and response to treatment with naltrexone. A secondary aim of this study is to examine the role of the Asp40 allele in alternating the subjective effects from alcohol use in alcohol dependent individuals that have been demonstrated in human laboratory experiments.

We hypothesize that naltrexone - but not placebo - will produce a greater clinical response during the 12 weeks of the trial in subjects with one or two copies of the Asp40 variant ("Asp40 positives") than in subjects homozygous for the Asn40 allele. Response to naltrexone will be measured by a reduction in the number of heavy drinking days (as defined by >5 drinks/day for males; >4 for females) during the 12 weeks of the trial.

We also expect that there will be an interaction between medication and genotype such that, as compared to the groups on placebo or homozygous for Asn40, Asp40 positive subjects randomized to naltrexone will report less "high" from alcohol consumption (on the Biphasic Alcohol Effects Scale), and the lowest levels of alcohol craving over time (on the Penn Alcohol Craving Scale).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female, 18 years of age or older, and of European or Asian descent.
2. Participant has a current DSM-IV diagnosis of alcohol dependence using the SCID/MINI.
3. The participant has signed a witnessed informed consent form.
4. Participant meets the following drinking criteria as measured by the Timeline Follow Back (TLFB): a. Drinks at least an average of 21 drinks/wk in the 60-day period prior to intake and b. Has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males, 4 or more in females) in this same pre-treatment period.
5. Participant has at least 48 hours of abstinence, as determined by subject report and breathalyzer measure immediately prior to randomization.
6. Participant scores below 8 on the Clinical Inventory of Withdrawal from Alcohol (CIWA) prior to starting Naltrexone.
7. Participant has adequate vision, hearing and ability to communicate to allow study participation.
8. Participant is able to speak, print and understand English.

Exclusion Criteria:

1. Participant meets DSM-IV criteria for dependence on any substance other than alcohol or nicotine in the last 6 months.
2. Participant has tested positive on the urine drug screen for opioids, benzodiazepines, or cocaine at the screening visit. Presence of THC is allowable.
3. Participant has a current or lifetime DSM-IV diagnosis of bipolar affective disorder, schizophrenia, or any psychotic disorder.
4. Participant has presence of unstable or serious medical illness such as a recent stroke, idiopathic seizure disorder, or cardiac disease.
5. Participant has severe liver disease (SGPT (ALT) or SGOT (AST) of at least 3 times normal value at the time of randomization or an elevated Total Bilirubin level without evidence of Gilbert's Syndrome.
6. Participant has taken any psychotropic medications (including disulfiram) regularly within the last seven days (14 for fluoxetine) prior to randomization or needs immediate treatment with a psychotropic medication (antidepressant, antipsychotic, benzodiazepine, or mood stabilizing medication). EXCEPTIONS: Zolpidem and ramelteon used sparingly if necessary for sleep; Oxazepam for alcohol detoxification; Seizure disorder medications.
7. Participant is over the age of 64 and has evidence of severe cognitive impairment as evidenced by a Mini-mental status exam (MMSE) score < 24.
8. Participant meets DSM-IV criteria for current major depression (non-substance induced), PTSD, or panic disorder.
9. Participant has suicidal or homicidal ideation necessitating inpatient hospitalization.
10. Participant is a pre-menopausal female who is pregnant, nursing, or not using a reliable method of contraception.
11. Participant is over age 64 and has evidence of severe cognitive impairment as evidenced by a Mini-mental status exam (MMSE) score less than 20.12. Participant is of African descent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2009-01-05 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2014-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oslin, MD, Principal Investigator — University of Pennsylvania/ Philadelphia VA Medical Center
Locations (4):
- United States (4):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oslin DW, Leong SH, Lynch KG, Berrettini W, O'Brien CP, Gordon AJ, Rukstalis M. Naltrexone vs Placebo for the Treatment of Alcohol Dependence: A Randomized Clinical Trial. JAMA Psychiatry. 2015 May;72(5):430-7. doi: 10.1001/jamapsychiatry.2014.3053. PMID 25760804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A sample of participants was recruited through advertisements in local media, referrals from physicians, or self-referrals. Recruitment occurred between January 2009 and September 2013. Participants were recruited from 5 sites.
Groups:
- Naltrexone Group ASP 40 Group: 50mg/day of naltrexone and ASP 40 carrier
- Placebo Group ASP 40 Group: Placebo group and ASP 40 carrier
- Naltrexone Group ASN 40 Group: Naltrexone 50mg/day and ASN 40 carrier
- Placebo Group ASN 40 Group: Placebo plus ASN 40 Carrier
Period: Overall Study
Arm/Group | Naltrexone Group ASP 40 Group | Placebo Group ASP 40 Group | Naltrexone Group ASN 40 Group | Placebo Group ASN 40 Group
Started | 38 | 44 | 73 | 66
Completed | 30 | 37 | 63 | 56
Not Completed | 8 | 7 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone Group ASP 40 Group | Placebo Group ASP 40 Group | Naltrexone Group ASN 40 Group | Placebo Group ASN 40 Group | Total
Number analyzed (Participants) | 38 | 44 | 73 | 66 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (13.4) | 46.9 (11.8) | 51.2 (13.0) | 48.2 (11.9) | 48.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10 | 11 | 31
  Male | 34 | 38 | 63 | 55 | 190
% Days Heavy Drinking [Mean (Standard Deviation); unit: % days of heavy drinking] | 68 (29.8) | 72.5 (27.8) | 67.5 (26.8) | 70.9 (28) | 69.9 (27.4)
% Days Drinking [Mean (Standard Deviation); unit: % days of any drinking] | 78.9 (23.1) | 82.7 (20.9) | 82.8 (20.2) | 82.5 (19.8) | 81.9 (20.7)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Naltrexone, as Measured by a Reduction in the Percent Days of Heavy Drinking Days (as Defined by >5 Drinks/Day for Males; >4 for Females) During the 12 Weeks of the Trial.
Time Frame: 12 weeks
Population: Repeated weekly measures of drinking outcomes were compared using generalized estimating equation models (GEE). The explanatory variables of primary interest comprised binary indicators for intervention group, genotype, and their interaction, a linear trend for time, and terms for interactions involving time and the group and genotype factors.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Naltrexone Group ASP 40 Group | Placebo Group ASP 40 Group | Naltrexone Group ASN 40 Group | Placebo Group ASN 40 Group
Number analyzed (Participants) | 38 | 44 | 73 | 66
percentage of heavy drinking days | 18.9 (21.7) | 17.9 (21.8) | 14.5 (19.0) | 21.7 (25.7)
Statistical Analysis 1: Comparison: Naltrexone Group ASP 40 Group vs Placebo Group ASP 40 Group vs Naltrexone Group ASN 40 Group vs Placebo Group ASN 40 Group; Test type: Superiority or Other; p = 0.32, Generalized Estimating Equation

ADVERSE EVENTS:
Time Frame: Adverse events were ascertained weekly.
Description: AE's were only counted if reported at a level of moderate to severe by patient self report.
Arm/Group | Naltrexone Group ASP 40 Group | Placebo Group ASP 40 Group | Naltrexone Group ASN 40 Group | Placebo Group ASN 40 Group
Serious Adverse Events (participants affected / at risk) | 0/38 | 2/44 | 1/73 | 2/66
Other Adverse Events (participants affected / at risk) | 1/38 | 2/44 | 4/73 | 3/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone Group ASP 40 Group (N=38) | Placebo Group ASP 40 Group (N=44) | Naltrexone Group ASN 40 Group (N=73) | Placebo Group ASN 40 Group (N=66)
inpatient detoxification (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitlized (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Diabetes
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone Group ASP 40 Group (N=38) | Placebo Group ASP 40 Group (N=44) | Naltrexone Group ASN 40 Group (N=73) | Placebo Group ASN 40 Group (N=66)
GI complaints (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — worsening pain
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Change in libido (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
While the study did not achieve the intended sample size, it is highly unlikely that a larger sample would have resulted in the demonstration of the expected moderating effect of the Asp40 allele.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No